CLINICAL TRIAL: NCT04691518
Title: Effect of Acute Intermittent Hypoxia in Healthy Individuals
Brief Title: Effect of Intermittent Hypoxia in Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Zev Rymer, Director Sensory Motor Performance Program, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00202448
Record Dates: First submitted 2020-12-22; First posted 2020-12-31 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: Acute Intermittent Hypoxia

STUDY DESIGN:
Intervention Model Description: Participants will participate in any of the interventions
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to Treatment or Placebo treatment when applicable
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Intermittent Hypoxia (AIH) (Active Comparator): Undergoing Acute Intermittent Hypoxia sessions
  Interventions: Other: Acute Intermittent Hypoxia
- Sham AIH (Placebo Comparator): Undergoing Sham AIH sessions
  Interventions: Other: Sham Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — 30 minute session of Acute Intermittent Hypoxia
  Arms: Acute Intermittent Hypoxia (AIH)
Other: Sham Acute Intermittent Hypoxia — 30 minute session of Sham Acute Intermittent Hypoxia
  Arms: Sham AIH

SUMMARY:
The use of acute intermittent hypoxia (AIH) has been examined in animal and human studies to gain an understanding of its effect on spinal excitability and synaptic strength. Subsequently, the investigators have learned that the use of AIH results in new protein formation and spinal plasticity. The use of acute intermittent hypoxia demonstrates a potential for therapeutic utilization in individuals with neurologic injuries. However, little is known about the effect of AIH in healthy individuals. This work is necessary to understand the mechanisms of AIH-induced plasticity. As such, this research study seeks to evaluate the impact of a single session AIH on upper extremity motor function in healthy individuals.

DETAILED DESCRIPTION:
The use of acute intermittent hypoxia (AIH), has been demonstrated, through human and animal studies, to be an effective way of increasing spinal motor excitability and strengthening residual synaptic connectivity. AIH utilizes short duration (<2 min) exposures to reduced oxygen levels (~10% inspired oxygen), with alternating exposures to air with normal oxygen levels (~21% inspired oxygen).

Previous publications demonstrate that AIH is a safe and effective intervention to modify motor function in individual with chronic incomplete spinal cord injuries. The use of AIH has been shown to influence the activation in musculature, within 60-120 minutes of administration. In addition, when coupling AIH with overground gait training, an increase in functional endurance, as evaluated through the 6 minute walk test, and gait speed, as evaluated through the 10 meter walk test, were demonstrated. In addition, the use of hypoxic training has been studied in healthy individuals and athletes; however, literature examining the effect of a single bout of AIH on performance is limited.

Although AIH has proven to be a promising treatment in enhancing spinal excitability and strengthening existing synaptic connections within individuals with chronic spinal cord injuries, further examination also needs to be made on the impact of AIH on motor function in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* No history of neurologic injury or progressive neuromuscular disorder
* Individuals ages 18-70 years old
* Must be medically stable with no history of cardiovascular instability, congestive heart failure or stroke
* Not currently (>2 weeks) on any medications related to spasticity
* No history of Sleep apnea
* Not a current smoker
* Able to comply with protocol/study requirements

Exclusion Criteria:

* Recent change in the use of narcotic, anti-inflammatory or pain medication
* unstable medical conditions or any other clinical observation that may affect the candidate's performance, health, safety or the ability to participate in the study determined by the treating therapist or coordinating staff
* Active participation in another movement research study or therapy program
* Anti-spasticity drug injection less than 3 months prior to beginning treatment
* Musculoskeletal pain that interferes with participation in study
* Women who are currently, may be, or planning on becoming pregnant
* for fMRI participation, participants will be excluded if they have:
* Metal fragments in eyes or face
* Implantation of any electronic devices such as (but not limited to) cardiac pacemakers, cardiac defibrillators, cochlea implants, or nerve stimulators
* Vascular surgery
* Claustrophobia
* Body piercing or tattoos

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-11-16 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Grip Strength | Immediately after acute intermittent hypoxia administration
  Change in strength from before acute Intermittent hypoxia to after administration

OTHER OUTCOMES:
Change in fMRI | Immediately after acute intermittent hypoxia administration
  fMRI evaluating changes in blood flow before and after acute intermittent hypoxia administration

CONTACTS AND LOCATIONS:
Overall Officials: William Rymer, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No